CLINICAL TRIAL: NCT02849392
Title: Effects of Pistachio Consumption on Body Composition, Blood Lipids, Bone Density, Satiety, Inflammatory Markers, and Erythrocyte Membrane Incorporation of Fatty Acids (The Cal Polys Pistachio Study)
Brief Title: Effects of Pistachio Consumption on Body Composition and Blood and Bone Indicators
Acronym: CPsPistachio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State Polytechnic University, Pomona (Other)
Collaborators: California Polytechnic State University-San Luis Obispo (Other); California State University Agricultural Research Institute (ARI) (Other); American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Dr. Bonny Burns-Whitmore, RD, Full Tenured Professor of Nutrition/Graduate Coordinator, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 002940-CPP Foundation; 082012-CPSLO ARI (Other Grant/Funding Number: California Agriculture Research Institute); 002940-CPP Foundation (Other Grant/Funding Number: American Pistachio Growers)
Record Dates: First submitted 2016-07-25; First posted 2016-07-29 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Pistachio; Body composition; Erythrocyte membrane incorporation of fatty acids; Dietary quality/micronutrient quality; Blood lipids; Inflammatory markers; Bone density; Bone turnover markers; Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pistachio (Experimental): Pistachio added 20% of kcals to diet
  Interventions: Other: Pistachio added 20% of kcals to diet
- No Pistachio (No Intervention): No pistachios in diet (control)

INTERVENTIONS:
Other: Pistachio added 20% of kcals to diet — Pistachio added 20% of kcals to diet
  Arms: Pistachio

SUMMARY:
Research investigating beneficial effects of regular pistachio feedings on body composition (BC) and blood lipids are limited, and there are no studies that have investigated the effects of feeding pistachios on bone density or membrane incorporation of fats. The purpose of this study is to examine the effects of pistachio consumption on body composition, bone density, markers of bone turnover, erythrocyte membrane incorporation of fatty acids, lipid status, inflammatory markers, dietary quality/micronutrients and satiety using a cross-over study with two 12-week treatment periods (pistachio added (20 percent of kcals) and a no-pistachio control diet), separated by 15-week washout period. The investigators will recruit 30 female students from Cal Poly, San Luis Obispo (CP-SLO) and female 30 students from Cal Poly, Pomona (CP-P) facilitating a collaborative project and using the expertise of both Dr. Laura Hall (CP-SLO) and Dr. Bonny Burns-Whitmore (CP-P). The investigators hope to show the health benefits of pistachios as part of an overall healthy lifestyle.

DETAILED DESCRIPTION:
Primary Research Objectives:

1. To examine the effects of a diet rich in pistachios on body composition
2. Examine incorporation of healthy fats into red blood cell (RBC) membranes
3. Determine changes in blood lipids, inflammatory markers and markers of bone turnover with pistachio consumption
4. Assess diet quality/micronutrient quality and satiety with pistachio consumption

Methods Investigators will employ a crossover design with two 12-week treatment periods (pistachio added and a no-pistachio control diet), separated by 15-week washout period, with 30 healthy students at each campus.

Subjects Female students enrolled at CP-SLO and CP-P will be invited to participate in the study. The first 30 qualified females will be enrolled in the study at each site. A screening questionnaire will determine eligibility. The interview will take ~5 minutes. This sample size provides more than adequate power (80%) to detect individual changes.

Recruitment Female students enrolled at CP-SLO and CP-P will be invited to participate in the study. Potential subjects will be notified by flyers, emails, adds on marquees, and peer recruitment in summer school classes. The information on the flyer and emails will be approved by the Institutional Review Boards and contain information regarding inclusion/exclusion criteria, length of study, and the risks and benefits. Participants will be asked to contact either Dr. Laura Hall (CP-SLO) or Dr. Bonny Burns-Whitmore (CP-P) and then potential participants will be asked to fill out a screening questionnaire to determine eligibility.

Study Design & Methods We will employ a randomized crossover design with two 12-week treatment periods: pistachio added (20% of kcals) and a no-pistachio control diet), separated by 15-week washout period, with 30 healthy female students at each campus. The first treatment period will be in Fall 2012 and the second treatment period will be in Spring 2013.

Randomization to treatment (pistachios) or habitual (control) diet and 24-hour recalls Randomization will be done utilizing a www.randomization.com list of random appointments to either the treatment group first or the control group first.

Materials and Procedures:

Study visits: Participants will come to the CP-SLO (n=30) or CP-P (n=30) site once a week during Fall quarter for 12 weeks and again during Spring quarter for 12 weeks to pick up their pre-measured pistachios for a total of 24 total study visits. At the initial visit, half the participants will be given pistachios to include in their diet as snacks or in meals (20 percent of kcals; intervention group) while half will continue their normal diets (control group). During, Spring, the other half of the participants will switch and consume the pistachios while the first half will not. Diet counseling will also be given at these visits and compliance to study protocols will be evaluated by counting the number of pistachio packages and looking at the participant's Unusual Diet Diary. At baseline and end of each treatment period, participants will have their height, weight, waist circumference, hip circumference, body composition measured and blood drawn at both sites. At CP-SLO they will also have their bone density measured (DXA). At the CP-P site they will have a fatty acid analysis performed to examine monounsaturated fatty acid incorporation into red blood cells (RBCs).

Calculation/Distribution of Pistachios and Initial/Weekly Study Visits During the lead-in period participants will meet initially and will be trained on keeping their food records by a Registered Dietitian (RD). During this week they will each keep a 3-day food record and turn it in immediately. The researchers will calculate how many pistachios each participant needs based off of the initial 3-day food record. This amount will be substituted as 20 percent of their usual caloric need and it will be pre-measured into daily individually-wrapped servings. The researches will meet with the participants weekly to give them a week's supply of their pre-measured packet of pistachios (one for each day). They will be asked to bring in their used wrappers to the weekly counseling meetings. At the weekly counseling meetings, participants will be shown how to incorporate the pistachios into their diet (either as snacks or in recipes) in an isocaloric diet, to check the participant's unusual diet diary and food records for accuracy, to review the 'MyPlate' guidelines and to check the empty pistachio wrappers for compliance. Participants will also get email/text reminders about meetings and reminder instructions on how to prepare for study visits.

Data Collected at both sites during Fall 2012 (wk 1 and wk 12) & Spring 2013 (wk 1 and wk 12):

Anthropometric Measurements: Body weight will be measured using a calibrated scale and recorded to the nearest 0.1 kg. Height will be measured using a stadiometer and recorded to the nearest 0.1 cm. Body mass index (BMI) will be calculated as weight (kg) divided by height (m) squared. Waist circumference will be measured using a flexible measuring tape between the middle of the bottom rib and iliac crest (top of the hip bone) and recorded to the nearest 0.1 cm. Hip circumference will be measured using a flexible measuring tape around the largest part of the hips (i.e. buttocks) and recorded to the nearest 0.1 cm. Measurements will be taken twice and averaged. We will also calculate their waist-to-hip ratio. Protocols will be based on NHANES III standardized procedures and student volunteers will be thoroughly trained on these protocols (see link-NHANES) Blood Pressure: Blood pressure will be taken using an automatic blood pressure monitor. Protocol will be based on Mayo Clinic standardized procedures and student volunteers will be thoroughly trained on these protocols (see link-Mayo Clinic).

Body Composition Measurement: Body fat percentage will be assessed by bioelectrical impedance analysis using the Tanita Body Composition Analyzer Scale (model TBF-310); from Tanita Corporation, (Tokyo, Japan). It will also be used to measure weight, body mass index (BMI), percent body fat, impedance, fat mass (TBF), fat free mass (FFM), total body mass (TBM), and total body water (TBW). The participants will need to fast for 12 hours before their study visit (i.e. no caffeine in the morning but 1.5 cups of water prior to the visit will be encouraged).

Food Records/Unusual Diet Diary (ie. Dietary Adherence & Compliance): Adherence and compliance to the assigned diets will be assessed using an Unusual Diet Diary (developed at CP-P), which is filled out by the participant when unusual quantities of foods or accidental pistachio consumption occurs, medical treatment is required, a suspected allergic reaction/side effect occurs or pharmaceuticals are consumed. If a participant experiences an allergic reaction to pistachios they will have been told to call 911 and after contacting the researchers, they will be removed from the study to limit further risk. Food records will be administered during each treatment to obtain information regarding the subject's diet and determine if the subject is adhering to treatment protocols. Participants will be thoroughly trained on how to keep accurate food records. Participants will be asked to perform 9 randomly selected food records throughout the study. Investigators will use the Nutrition Data System for Research (NDSR) from the University of Minnesota on both campuses for the diet analysis software (see NDSR link).

Satiety and Hunger ratings: Participants will rate their hunger using a rating scale (1-10) before, during and after each snack or meal directly on their 9 required food records during each treatment, and will use a validated visual analog scale (VAS) to rate their hunger after consuming their snack or meal with pistachios for the intervention group and randomly chosen snacks/meals for the control group. Participants will be given binders with the food record forms and VAS questionnaires in them with the randomly chosen dates and instructions listed. Completed forms will be checked for accuracy and collected at the weekly visits from the binders.

Physical Activity Questionnaire: Participants will be asked to recall their physical activity level over the preceding week (7 day recall) using the 2002 International Physical Activity Questionnaire (IPAQ) short form. Participants will be encouraged to maintain their usual levels of physical activity.

Chem Panel/Iron Panel/Blood Lipids: Blood will be drawn on campus at the Health Center at week 1 and 12 to examine a lipid panel, a standard chem. panel and iron status. The participants will need to fast for 12 hours before the blood draw, however, consuming 1.5 cups of water in the morning will be encouraged.

Inflammatory Markers: Blood will be drawn on campus at the Health Center at week 1 and 12 to examine inflammatory markers (ie, C-reactive protein (CRP), tumor necrosis factor alpha (TNFa), and interleukin-6 (IL-6)). The participants will need to fast for 12 hours before the blood draw, however, consuming 1.5 cups of water in the morning will be encouraged.

Markers of Bone Turnover: Blood will be drawn on campus at the Health Center at week 1 and 12 to examine markers of bone turnover.

Data Collected at the Cal Poly, SLO site only :

Body Composition/Bone Mineral Density (DXA): Full-body DXA (iDXA, General Electric Healthcare) will be used to determine body fat mass, body fat percentages, lean body mass and bone mineral density of each subject. A pregnancy test will be given to participants before the test to ensure safety of the fetus. If positive, the participant will be asked to terminate their participation in the study.

Data Collected at the Cal Poly, Pomona site only:

Erythrocyte Membrane Incorporation (Lipomics): Erythrocytes membranes will be measured for all fatty acids. Erythrocytes will be packed in dry ice and shipped overnight to Lipomics Technologies, West Sacramento, California 95691.

Data Analysis: A statistician will be consulted and all statistical analyses will be conducted using Statistical Analysis Software (SAS version 9.2). Time-repeated analysis of variance (ANOVA) will be performed for comparisons between the variables during the two time points and ANOVA's will be performed between the two treatment groups. Spearman's correlation will be used to examine associations between the variables.

Debriefing of Participants: Subjects will be consented to this study and will be aware of the purpose of this study. All subjects will be given a copy of the consent form.

Results Dissemination Plan

The dissemination plan for the results of this project includes but is not limited to:

* Publication in peer-reviewed journals (i.e. Journal of Nutrition, The Journal of Clinical Nutrition, The Journal of the Academy of Nutrition and Dietetics (AND), the American Journal of Public Health, Journal of Family and Consumer Science).
* Publication in newsletter articles and research bulletins
* Publication on the Cal Poly Pomona web site, Agriscapes, e-mail announcements, presentation at poster sessions
* Presentation at scientific meetings (i.e. Experimental Biology).

ELIGIBILITY:
Inclusion Criteria:

* Cal Poly, SLO or Pomona biological female students (Age 18-40 yrs, BMI 18.5-25).
* Must like eating pistachios.
* Free of chronic diseases.

Exclusion Criteria:

* Non-Cal Poly students and males.
* Allergies to pistachios or other nuts.
* Eat excessive amounts of nuts.
* Less than 18 yrs old or older than 40 yrs.
* Female BMI less than 18.5 or greater than 25.
* Any disease or underlying condition that requires treatment that may affect metabolism, normal dietary intake or physical activity levels.
* Use of medications that affect fat malabsorption, use of laxatives, liver disease, kidney disease, thyroid disease, Diabetes, hypertension, dyslipidemia, or pregnancy, cancer.
* Pacemakers or metal pins or plates in the body
* Unwillingness to follow study protocol
* Must avoid eating other nuts, fish oil and flax seed/oil.
* Any chronic disease.
* Excessive consumption of alcohol.
* Elite Athletes will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition as measured with the Tanita scale TBF-310 at week 12 as compared to change in body composition from baseline with inclusion of 20% Kcals from pistachios measured at week 12. | 24 weeks-12 weeks intervention, 12 weeks no intervention
  Changes in body composition will be determined by the Tanita scale and/or by DXA differences from baseline to end in the pistachio intervention as compared to not consuming 20% Kcals of pistachios for 12 weeks

SECONDARY OUTCOMES:
Change from baseline in RBC membrane fatty acids as measured by Lipomics technology at week 12 as compared to change in RBC membranes from baseline to 12 weeks when consuming 20% of diet kcals from pistachios. | 24 weeks-12 weeks intervention, 12 weeks no intervention
  Using Lipomics laboratory patented technology (Metabolomics now) they will determine the fatty acid incorporation into red blood cell (RBC) membranes differences from baseline to end in the pistachio intervention as compared to not consuming pistachios for 12 weeks

OTHER OUTCOMES:
Change from baseline in blood lipids, inflammatory and bone markers as measured by a contracted laboratory at week 12 as compared to change from baseline to week 12 when consuming 20% of diet kcals from pistachios. | 24 weeks-12 weeks intervention, 12 weeks no intervention
Change in diet quality as measured by the NDS-R Software during the diet record keeping periods (3 times each arm for 3 days) during the 12 weeks for 20% dietary Kcals from pistachios and for the no-pistachio treatment arm. | 24 weeks-12 weeks intervention, 12 weeks no intervention
  The NDS-R Software is produced by the University of Minnesota Reagants. Diets were randomized for each participant 3 times for 3 days each during each of the 12 week arms. This resulted in 18 total diet records for each participant.
Change in satiety as measured by the Visual Analog Scales (VAS) during the diet record keeping periods (3 times each arm for 3 days) during the 12 weeks for 20% dietary Kcals from pistachios and for the no-pistachio treatment arm. | 24 weeks-12 weeks intervention, 12 weeks no intervention
  Diets were randomized for each participant 3 times for 3 days each during each of the 12 week arms, and the VAS satiety questionnaire was used to measure satiety when pistachios were consumed or at a randomized meal if the participant was not consuming pistachios in that treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Oates, MD, Study Director — California Polytechnic University-San Luis Obispo

IPD SHARING:
Plan to Share IPD: Yes
lipid and blood data

REFERENCES:
- See also: MAYO CLINIC — http://www.mayoclinic.com/health/how-to-measure-blood-pressure/MM00785/
- See also: NDS-R Software — http://www.ncc.umn.edu/products/